CLINICAL TRIAL: NCT06392126
Title: An Open-label Study of an Experimental Antisense Oligonucleotide Treatment for a Single Participant With Amyotrophic Lateral Sclerosis (ALS) Due to a Pathogenic Variant in CHCHD10
Brief Title: Personalized Antisense Oligonucleotide Therapy for A Single Participant With CHCHD10 ALS
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-011476
Record Dates: First submitted 2024-04-24; First posted 2024-04-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-CHCHD-001

INTERVENTIONS:
Drug: nL-CHCHD-001 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with amyotrophic lateral sclerosis (ALS) due to a pathogenic variant in CHCHD10

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with amyotrophic lateral sclerosis (ALS) due to a pathogenic variant in CHCHD10

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s).
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.
* Genetically confirmed neurological disorder.

Exclusion Criteria:

* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures.
* Use of an investigational medication within less than 5 half-lives of the drug at enrollment

Min Age: 48 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R).
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on ALS Cognitive Behavioral Screen (ALS-CBS)
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Amyotrophic Lateral Sclerosis Assessment Questionnaire 5 (ALSAQ-5).
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on vital capacity performance.
Disease biomarkers | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in serum/plasma and CSF neurofilament light chain levels
Survival | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in survival status

SECONDARY OUTCOMES:
Safety and tolerability | Baseline to 12 months
  Incidence and severity of adverse events
Safety and tolerability | Baseline to 12 months
  Emergent abnormalities in physical exam
Safety and tolerability | Baseline to 12 months
  Emergent abnormalities in neurological exam
Safety and tolerability | Baseline to 12 months
  Emergent abnormalities in safety labs (CSF, chemistry, hematology, coagulation, and urinalysis)

CONTACTS AND LOCATIONS:
Overall Officials: Björn E. Oskarsson, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No